CLINICAL TRIAL: NCT01077531
Title: A Randomized, Placebo-controlled, Single-blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of Otelixizumab in Rheumatoid Arthritis Subjects
Brief Title: Safety, Pharmacodynamics and Pharmacokinetics of GSK2136525 Repeat Dose in Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The risk-benefit ratio for patients has changed since we initiated the study, and that the study in its current form cannot be justified
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111601
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; intravenous infusion; long-term followup
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — otelixizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Otelixizumab (Active Comparator): Otelixizumab (GSK2136525) is a humanised, aglycosyl, non-mitogenic, anti CD3 monoclonal antibody (MAb).
  Interventions: Drug: Otelixizumab
- Placebo (Placebo Comparator): Matching placebo for intravenous infusion
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Otelixizumab — Otelixizumab injection for intravenous infusion. Otelixizumab (GSK2136525) is a humanised, aglycosyl, non-mitogenic, anti CD3 monoclonal antibody (MAb).
  Arms: Otelixizumab
Drug: Matching placebo — Matching placebo for intravenous infusion
  Arms: Placebo

SUMMARY:
The assessment of otelixizumab in rheumatoid arthritis subjects will provide safety, tolerability, pharmacodynamic and pharmacokinetic information which will enable the identification of appropriate safe and well-tolerated dosage regimens to be used in clinical efficacy studies. This study will consist of a screening phase, followed by a treatment period where four cohorts of subjects will receive 5 daily intravenous infusions of otelixizumab. The cumulative dose will increase in each successive cohort and infusion rates can be adjusted based on signs and symptoms of cytokine release syndrome and to ensure the specified maximum infusion rate is not exceeded. Serial blood samples will be obtained for clinical laboratory testing, determination of pharmacodynamic markers, serum otelixizumab PK parameters, exploratory biomarkers and immunogenicity. Safety and pharmacodynamic data from the previous cohort(s) will be evaluated prior to dosing subsequent cohorts to ensure safety. Adverse events, laboratory values, vital signs and ECG's will be monitored closely during this study. All subjects in the study will undergo long-term follow-up out to 48 months to monitor patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 75 years of age inclusive.
* Female subjects of: a. non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 mIU/ml and estradiol <40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method. b. Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 of the protocol for an appropriate period of time to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for at least 2 weeks prior to dosing and for at least 60 days after the last dose.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1 of the protocol. This criterion must be followed from the time of the first dose of study medication until at least 60 days after the last dose.
* Body mass index within the range 18.5 - 35 kg/m2 inclusive.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form and willing and able to follow the procedures outlined in the protocol.
* A 12-lead ECG at pre-study screening measured in triplicate, which in the opinion of the Principal Investigator or physician designee has no abnormalities that will compromise safety in this study. QTcB < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
* The subject has a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology.
* The subject tests positive for Rheumatoid factor.
* The subject has active disease with at least 3 swollen and 3 tender joints, early morning joint stiffness ≥ 30 minutes and a serum CRP>5mg/L (3 out of 4) at screening.
* The subject has ACR functional class I-III.
* The subject has persistent disease activity in spite of therapy with at least one DMARD.
* The subject has not previously received otelixizumab or any other anti-CD3 monoclonal antibody, e.g., OKT3 (muromonab or Orthoclone), ChAglyCD3, or hOKT3γ1 (ala ala), and is willing to refrain from using any such antibody for 2 years after the last dose of study drug unless invited to participate in possible future studies with otelixizumab.
* If taking methotrexate, the patient must have been taking methotrexate for at least 12 weeks and to be on a stable dose of methotrexate (7.5-25 mg/week) for at least four weeks prior to dosing and be willing to remain on this up to 12 weeks after last dose of the investigational product in this study unless change required for clinical management of disease activity or safety.
* If sulfasalazine is being taken, the patient must have been taking sulfasalazine for at least 12 weeks and to be on a stable dose within local treatment guidelines for at least 4 weeks prior to dosing and be willing to remain on this dose for at least 12 weeks after the last dose of study drug unless change required for clinical management of disease activity or safety.
* If leflunomide is being taken, the patient must have been receiving this DMARD for at least 6 months prior to dosing with otelixizumab and the DMARD dose has been stable dose within local treatment guidelines for 12 weeks prior to dosing with study drug.
* Patients on glucocorticoids e.g. prednisolone (≤10mg/day), must be on stable dosing regimens for at least 4 weeks prior to dosing and be willing to remain on this regime for at least 12 weeks after the last dose of study drug.
* PRN use is acceptable for NSAIDS and COX-2 inhibitors within local treatment guidelines.
* The subject is seropositive for EBV with <10,000 copies of EBV DNA per 106 lymphocytes (qPCR) or seronegative with no evidence of acute EBV infection (asymptomatic, negative EBV IgM and EBV viral load of <10,000 per 106 lymphocytes).
* The subject has no current or prior malignancy, other than non-melanoma skin cancer (subject must have had fewer than 5 occurrences of non-melanoma skin cancer, and the last occurrence must not be within 3 months of study entry).

Exclusion Criteria:

* Subjects with a history of significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis, or Felty's syndrome).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening; current or chronic history of liver disease.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* A positive EIA test for syphilis.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) or planning to take any investigational drug for the planned duration of study participation (6 months after the last dose of study drug).
* Previous or current exposure to biologic cell-depleting anti-rheumatic therapies, including investigational compounds (e.g. anti-CD11a, anti-CD-20, anti-CD22, anti-BLyS/BAFF, anti-CD3, anti-CD5, anti-CD52).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive (serum or urine) hCG test at screening or prior to dosing, or lactating females.
* The subject is currently receiving or has received an anti-rheumatic biological therapy within the following specified periods prior to dosing: Within 4 weeks: Glucocorticoid unless given in doses equivalent to ≤10 mg of prednisolone/day; Intramuscular. or i.v. corticosteroids; Live/attenuated vaccinations; Cyclosporine; Etanercept, within 8 weeks: Rituximab; Infliximab; Adalimumab or other subcutaneous anti-TNF/TNF-Rc therapy; Anakinra; Abatacept; Tocilizumab; Certolizumab, within 24 weeks: Anti-cancer therapy (e.g. alkylating agents, anti-metabolites, purine analogues, monoclonal antibodies).
* The subject has received immunization with a vaccine within 4 weeks before the first dose of study drug or requires a vaccine within 30 days after the last dose of study drug.
* A CD4+ lymphocyte count outside the range of 0.53 - 1.76 × 109/L during Screening.
* The subject has had a significant systemic infection during the 6 weeks before the first dose of study drug (e.g., infection requiring hospitalization, major surgery, or IV antibiotics to resolve); other infections, e.g., bronchitis, sinusitis, localized cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-by-case basis by the investigator regarding whether they are serious enough to warrant exclusion).
* The subject has received a course of oral antibiotics within 2 weeks of dosing day one.
* History of recurrent or chronic infection.
* The subject has had a splenectomy.
* Subjects with a screening chest X-ray suggestive of TB without documentation of adequate TB treatment will be excluded. Screening for latent TB infection using intradermal injection of tuberculin (e.g. the Mantoux test or equivalent) should be conducted in accordance with local guidelines. The tuberculin skin test results should be evaluated according to the criteria for immunocompromised subjects. Subjects with a positive skin tuberculin test should be excluded if the investigator judges the patient to be at risk of latent TB infection.
* The subject has undergone any major surgical procedure within the 8 weeks before signing the consent form, or planning to undergo any such surgery within the 3 months after the last dose of study drug.
* Has clinically significant cardiovascular and/or cerebrovascular disease including, but not limited to: Previous history of stroke or transient ischemic attack; Active, unstable coronary heart disease within the past 6 months; Documented myocardial infarction within a year of screening; Any cardiac surgery including percutaneous transluminal coronary angioplasty or coronary artery bypass graft surgery within a year prior to screening; Unstable angina; Clinically significant arrhythmia or valvular heart disease within the past year; Congestive heart failure with New York Heart Association Class II to Class IV symptoms. Class I is acceptable; Untreated hypertension, with systolic pressure greater than 160mm Hg and/or diastolic pressure greater than 95mm Hg.
* Predisposition to thromboembolic disease, or thromboembolic event (excluding superficial) in past 12 months.
* Uncontrolled medical conditions: Significant concurrent, uncontrolled medical condition including, but not limited to renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral psychiatric disease, or evidence of demyelinating disease.
* Positive plasma / white cell JC virus (JCV) PCR (either compartment).
* The subject has a condition or situation that, in the investigator's judgment, is likely to cause the subject to be unable or unwilling to participate in study procedures or to complete all scheduled assessments.
* The subject has clinically significant abnormal laboratory values during the Screening period, other than those due to RA. Abnormal values are permitted if, upon re-test, the abnormality was resolved (ALT <2xULN, AST <2xULN).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04-28 (Actual); Primary Completion 2013-03-19 (Actual); Study Completion 2013-03-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple doses of otelixizumab: adverse events, ECGs, laboratory safety results, Epstein-Barr Virous viral load, JCV detection. | 48 months
Saturation and modulation of CD3/TCR complex on peripheral blood T cells | Six months
Individual absolute and percentage circulating peripheral T lymphocytes and CD4+ and CD8+ subset counts | Six months

SECONDARY OUTCOMES:
Serum concentrations of otelixizumab and PK parameters | Five days
Individual absolute and percentage circulating Treg as measured by foxP3+ and CD4 + foxP3+ subsets | Six months
Anti-otelixizumab antibody titres and whether detected antibodies are neutralising | Three months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Yaroslavl
- Spain (2):
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
- United Kingdom (2):
  - GSK Investigational Site, Cambridge, Cambridgeshire
  - GSK Investigational Site, Newcastle, Northumberland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register